CLINICAL TRIAL: NCT02940548
Title: A Comparative Study for the Effects of Nifedipine GITS and Amlodipine Besylate on Recovery of Blood Pressure Rhythm and Arterial Stiffness in the Young and Middle-aged Subjects With Non-dipper Hypertension
Brief Title: Nifedipine GITS and Amlodipine Besylate on Recovery of Blood Pressure Rhythm and Arterial Stiffness
Acronym: NARRAS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The patient recruitment and follow-ups were influenced with the pandemic of COVID-19
Sponsor: Jing Liu (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Jing Liu, Chief Physician, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016PHB013-02
Record Dates: First submitted 2016-10-15; First posted 2016-10-21 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
Keywords: non-dipper hypertension; young; middle-aged; ambulatory blood pressure monitoring; arterial stiffness; nifedipine gastrointestinal therapeutic system (GITS)
MeSH Terms: conditions — Hypertension | interventions — Nifedipine; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nifedipine GITS (Active Comparator): Nifedipine GITS 30~60mg/day
  Interventions: Drug: Nifedipine GITS
- Amlodipine besylate (Active Comparator): Amlodipine besylate 5~10mg/day
  Interventions: Drug: Amlodipine besylate

INTERVENTIONS:
Drug: Nifedipine GITS — Nifedipine GITS 30~60mg/day for 8 weeks
  Other Names: Adalat
  Arms: Nifedipine GITS
Drug: Amlodipine besylate — Amlodipine besylate 5~10mg/day for 8 weeks
  Other Names: Norvasc
  Arms: Amlodipine besylate

SUMMARY:
This trial evaluates the effects of Nifedipine GITS and Amlodipine besylate on blood pressure rhythm restoration and arterial stiffness in young and middle-aged non-dipper hypertensives. Half of participants will receive Nifedipine GITS, half of half will take medicine in the morning or at night. While the other half participants will take amlodipine besylate, whom will also be assigned taking medicine in the morning or at night. Ambulatory blood pressure monitoring and arterial stiffness examination will be performed before and after pharmaceutical intervention.

DETAILED DESCRIPTION:
Written informed consent will obtained from all the participants. All the adverse reaction or adverse event, related or unrelated to the study drug, will be recorded in detail, including the occurrence time, symptoms and vital signs, degree, duration, laboratory test indexes, treatment methods and results, process, follow-up time, etc.

If serious adverse event occurs, study drugs should be stopped and necessary remedy should be delivered immediately. At the same time, the investigator must report it to the local drug supervision, medical ethics committee and China Food and Drug Administration.

-

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate (Office blood pressure : 140 mmHg =< systolic blood pressure (SBP) <180 mmHg and / or 90 mmHg =< diastolic blood pressure (DBP) <110 mmHg) , non-dipper (ambulatory blood pressure monitoring (ABPM): night-time mean SBP / day-time mean SBP >=0.9 and night-time mean SBP >=120 mmHg) hypertensive subjects, who is drug treatment-naive or previously treated but discontinued for 2 weeks or more
* The subject is voluntary to participate in the study and has signed the informed consent form

Exclusion Criteria:

* Known allergy to any component of Nifedipine and Amlodipine
* Office SBP >=180 mmHg and / or DBP >=110 mmHg in the screening period
* The patient who is taking calcium antagonists (monotherapy or combination with other drugs)
* Evidences of secondary hypertension
* History of cerebrovascular events, cardiac failure, serious coronary artery disease within 12 months
* Type 1 diabetes mellitus (DM)
* Severe liver diseases or renal insufficiency
* The pregnant woman, the woman who may be pregnant or plan to be pregnant, or the lactating woman
* The subject who needs to work at night (on night shift)
* Other reasons that the subject can not participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Nighttime systolic blood pressure reduction | 8 weeks
  Compare the effects of two active drugs on nighttime systolic blood pressure reduction

SECONDARY OUTCOMES:
The proportion of recovery of dipper rhythm of blood pressure | 8 weeks
  Compare the effects of two active drugs and different time administration on recovery of dipper rhythm. The proportion of blood pressure dipper rhythm at 8 weeks after two drugs administration will be calculated. The proportion of dipper rhythm at 8 weeks after two drugs administration in the morning or at night will also be calculated.
Change of pulse wave velocity | 8 weeks
  Compare the effects of two active drugs on pulse wave velocity(PWV). PWV will be measured before and after 8 weeks two active drugs administration.

OTHER OUTCOMES:
Incidence of treatment-related adverse events | 8 weeks
  change of heart rate; change of liver and kidney function; other adverse reactions, such as edema, flushing, etc during 8 weeks of intervention and follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de la Sierra A, Redon J, Banegas JR, Segura J, Parati G, Gorostidi M, de la Cruz JJ, Sobrino J, Llisterri JL, Alonso J, Vinyoles E, Pallares V, Sarria A, Aranda P, Ruilope LM; Spanish Society of Hypertension Ambulatory Blood Pressure Monitoring Registry Investigators. Prevalence and factors associated with circadian blood pressure patterns in hypertensive patients. Hypertension. 2009 Mar;53(3):466-72. doi: 10.1161/HYPERTENSIONAHA.108.124008. Epub 2009 Jan 26. PMID 19171788
- [Derived] Liu J. A comparative study for the effects of nifedipine GITS and amlodipine besylate administrated in daytime or at nighttime on recovery of blood pressure rhythm and arterial stiffness in the young and middle-aged subjects with non-dipper hypertension (NARRAS): Design and rationale. Int J Clin Pract. 2020 Dec;74(12):e13628. doi: 10.1111/ijcp.13628. Epub 2020 Sep 3. PMID 32726499